CLINICAL TRIAL: NCT03051074
Title: Examining the Effects of Reduced Environmental Stimulation on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Principal Investigator, Sahib Khalsa, Principal Investigator, Laureate Institute for Brain Research, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-002 Float-Anxiety
Record Dates: First submitted 2017-01-09; First posted 2017-02-13 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Generalized Anxiety Disorder; Agoraphobia; Panic Disorder; PostTraumatic Stress Disorder; Social Anxiety Disorder; Major Depressive Disorder
Keywords: Anxiety; Floating
MeSH Terms: conditions — Generalized Anxiety Disorder; Agoraphobia; Panic Disorder; Stress Disorders, Post-Traumatic; Phobia, Social; Depressive Disorder, Major; Anxiety Disorders | interventions — Divorce

STUDY DESIGN:
Intervention Model Description: On the 2nd session, participants will be randomly assigned to start in the pool condition or comparison condition. Following a 1-week washout period, they will crossover to the other condition.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Floating (Experimental): The participant will float supine in water with a high concentration of Epsom salt for up to 90 minutes on three separate occasions
  Interventions: Behavioral: Floating
- Comparison condition (Active Comparator): The participant will watch a relaxing 90 minute film as a comparison condition
  Interventions: Behavioral: Comparison

INTERVENTIONS:
Behavioral: Floating — Floating supine in a pool saturated with Epsom salt for up to 90 minutes
  Arms: Floating
Behavioral: Comparison — Watching a relaxing film for up to 90 minutes
  Arms: Comparison condition

SUMMARY:
The studies proposed in this protocol aim to explore the anxiolytic properties of floating as it relates to the central and autonomic nervous system.

DETAILED DESCRIPTION:
The human brain is constantly bombarded with sensory information from the external world. This series of studies aim to explore the effects of reducing environmental stimulation using specially designed floatation pools that minimize visual, auditory, tactile, proprioceptive, and thermal input to the brain. Previous research has shown that "floating" in this unique setting can significantly reduce levels of anxiety, stress, blood pressure, and cortisol, while significantly increasing levels of both subjective and physiological forms of relaxation. Much of this past research contained various methodological weaknesses, including small sample sizes and lack of a control condition. Moreover, very little is known about the potential benefits of floating in clinical populations, and essentially nothing is known about the effects of floating on the brain. The studies proposed in this protocol aim to further explore floating's potentially salubrious effect on the autonomic nervous system, while beginning to investigate its largely unknown effect on the central nervous system. The researchers have attempted to improve upon the weaknesses of past research by using larger sample sizes and a control condition. The current project is focused on documenting the subjective, physiological and neural effects of floating in healthy and anxious populations. The subjective effects of floating will be examined using self-report measures and the experience sampling method. The physiological effects of floating will be examined using waterproof and wireless tracking of blood pressure, heart rate, respiration, and movement, in addition to collecting measures of cortisol and magnesium. The neural effects of floating will be examined using waterproof and wireless EEG collected during the float experience, as well as using functional magnetic resonance imaging (fMRI) collected before and immediately after floating. An exteroceptive control condition aims to examine each participant's baseline physiological state while participants watch a neutral documentary film. This program of research constitutes the first systematic investigation of floating on the body and the brain, and the findings have the potential to illuminate the physiological and neural correlates of the relaxation response induced by the floating experience.

ELIGIBILITY:
Inclusion Criteria for anxious subjects:

1. Overall Anxiety Severity and Impairment Scale (OASIS) score ≥ 8
2. Anxiety Sensitivity Index 3 (ASI-3) score of ≥ 29
3. Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnosis of an anxiety disorder or PTSD as determined by the Mini International Neuropsychiatric Interview (MINI Version 6.0)
4. Comorbid conditions are acceptable (except those listed in the exclusion criteria).

Inclusion Criteria for healthy subjects:

1. Overall Anxiety Severity and Impairment Scale (OASIS) score < 4
2. Anxiety Sensitivity Index 3 (ASI-3) score < 13
3. No DSM-V diagnoses as determined by the Mini International Neuropsychiatric Interview (MINI Version 6.0) and no history of neurological or psychiatric issues.

Exclusion Criteria:

1. Has any of the following DSM-V disorders:

   1. Schizophrenia Spectrum and Other Psychotic Disorders
   2. Bipolar and Related Disorders
2. Is currently being treated for their psychiatric condition as an inpatient
3. Active suicidal ideation with intent or plan
4. Participant is morbidly obese (BMI > 40) or underweight (BMI < 17).
5. Certain drugs or medications consumed within the past week including any psychoactive drugs (e.g., MDMA, LSD, psilocybin, peyote, phencyclidine, ketamine). For all other medications, the participant will be required to be stably medicated prior to participation (defined as having taken the medication for 6 weeks or longer).
6. Participant has a history of unstable liver or renal insufficiency; glaucoma; diabetes; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
7. Pregnancy as detected by a urine test.
8. Non-correctable vision or hearing problems.
9. Unwillingness or inability to complete any of the major aspects of the study protocol. However, failing to complete some individual aspects will be acceptable (e.g., being unwilling to answer individual items on a questionnaire).
10. MRI contraindications including: cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/ wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60-120 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Spielberger State Anxiety Inventory (STAI-S) change score | The investigators will calculate the pre- to post-float change score following each session (up to 3 float sessions + 1 comparison session completed over a 1 year time period; each session will be spaced apart by a minimum of 7 days)
  A valid and reliable psychological inventory consisting of 20 self-report items pertaining to state anxiety. The investigators will calculate pre- to post-float change scores.

SECONDARY OUTCOMES:
Blood pressure changes during the float experience | These measures will be acquired during the 2nd float session and comparison session, with each session spaced apart by a minimum of 7 days
Heart rate variability changes during the float experience | These measures will be acquired during the 2nd and 3rd float sessions + comparison session completed over a 1 year time period, with each session spaced apart by a minimum of 7 days
EEG changes during the float experience | EEG will be acquired during the 2nd and 3rd float sessions + comparison session completed over a 1 year time period, with each session spaced apart by a minimum of 7 days
Brain activation and connectivity changes from pre- to post-float as measured with functional magnetic resonance imaging (fMRI) | fMRI will be acquired immediately before and after the 3rd float session (completed over a 1 day time period)
Bioassay changes in magnesium, sulfate, cortisol, and inflammatory markers | Samples will be acquired before and after the 2nd and 3rd float sessions + comparison session completed over a 1 year time period, with each session spaced apart by a minimum of 7 days
  Blood and urine samples
Subjective changes in emotion and mood | Self-report measures acquired before and after each session (3 float sessions + comparison session completed over a 1 year time period, with each session spaced apart by a minimum of 7 days)
  Examining pre- to post-float change scores on various self-report measures (e.g., PANAS-X)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Feinstein, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flux MC, Fine TH, Poplin T, Al Zoubi O, Schoenhals WA, Schettler J, Refai HH, Naegele J, Wohlrab C, Yeh HW, Lowry CA, Levine JC, Smith R, Khalsa SS, Feinstein JS. Exploring the acute cardiovascular effects of Floatation-REST. Front Neurosci. 2022 Dec 9;16:995594. doi: 10.3389/fnins.2022.995594. eCollection 2022. PMID 36570829
- [Derived] Feinstein JS, Khalsa SS, Yeh HW, Wohlrab C, Simmons WK, Stein MB, Paulus MP. Examining the short-term anxiolytic and antidepressant effect of Floatation-REST. PLoS One. 2018 Feb 2;13(2):e0190292. doi: 10.1371/journal.pone.0190292. eCollection 2018. PMID 29394251